CLINICAL TRIAL: NCT04553185
Title: Study on the Effects of Single Nucleotide Polymorphisms in Aquaporin-4 (AQP4) Gene on the Clinical Phenotype in Patients With Idiopathic and Familial Parkinson's Disease.
Brief Title: Aquaporin-4 Single Nucleotide Polymorphisms in Patients With Idiopathic and Familial Parkinson's Disease
Status: Active, not recruiting | Type: Observational
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Other Study IDs: 2020 21/02
Record Dates: First submitted 2020-08-26; First posted 2020-09-17 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; AQP4; Glymphatic System; Genetics
MeSH Terms: conditions — Parkinson Disease | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — A venous sample will be collected from all participants. The venous sample will serve for genetic testing for Single Nucleotide Polymorphisms in the Aquaporin-4 gene and genetic testing for mutations in the following Parkinson's disease-related genes SNCA, LRRK2, VPS35, PARK2, PINK1, DJ-1, SYNJ1, DNAJ6, FBXO7, PLA2G6, LRP10, GBA and MAPT in a cohort of PD patients, as well as for the determination in the blood of the levels of the following substances: α-synuclein (total and oligofragmented), S100β, LRP1, and ABCB1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Parkinson's disease patients: Patients with idiopathic or familial Parkinson's disease
  Interventions: Other: Study procedure

INTERVENTIONS:
Other: Study procedure — All participants will undergo a collection of demographic data, personal and family history for PD, a neurological examination and administration of clinical scales. All participants will undergo a collection of venous blood sample. At the end of the visit they will receive a wristwatch to monitor their sleep at home (Actigraph) and a sleep diary, together with a prepaid envelope to post the watch and the diary back to the investigators. They will also receive a link for a series of online tests for non-motor symptoms related to Parkinson's disease that they can complete remotely at home.

SUMMARY:
The purpose of this study is to understand the relationship between problems in sleep, genetic variations in the Aquaporin-4 gene (AQP4), and the development of Parkinson's Disease.

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is a progressive neurodegenerative disease characterized by the abnormal deposition in the brain of aggregates called Lewy Bodies, packed with a protein called α-synuclein. The mechanisms why this protein accumulates in the brain of patients with PD, as well as its relationship with clinical symptoms, is unknown.

Recently, an internal mechanism of drainage of waste proteins called glymphatic system has been identified and characterized. This system is silent during wakefulness and works during sleep. When it is active, a virtual space between the blood capillaries and cells of the brain called astrocytes opens and lets out waste products from the brain. This process is mediated by a protein of the astrocytes called Aquaporin-4 (AQP4). Preclinical studies have shown that the function of this system could be critical for the clearance of β-amyloid, a protein linked with the development of Alzheimer's Disease. Studies in humans have shown that genetic variations some parts of the AQP4 gene, defined as single nucleotide polymorphisms, may increase the likelihood to develop an aggressive form of Alzheimer's Disease. However, no studies in humans have ever been performed in Parkinson's disease and α-synuclein.

In this study, the investigators aim to elucidate whether genetic variations in the AQP4 gene contribute to variations in the clinical presentation and progression of sporadic and genetic forms of Parkinson's disease. To do so, the genetic profile of patients will be determined through a small venous blood sample collection. This will be coupled with clinical and sleep assessment.

ELIGIBILITY:
Inclusion Criteria:

* 18-85 years of age
* Able to give informed consent
* Able to perform online neuropsychological examinations
* Diagnosis of PD according to Brain Bank Criteria
* No presence or personal or family history of other neurological or psychiatric disorders

Exclusion Criteria:

* Presence of other neurological disorders and known intracranial co-morbidities such as stroke, haemorrhage, space-occupying lesions
* Inability to perform online neuropsychological assessment
* Inability to have access to informatics technology to perform the online assessment tests
* Inability to travel for the assessments
* Native language different from English

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of Parkinson's disease according to Published Criteria.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2018-11-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Association between genetic variations in the AQP4 gene and worse motor symptoms in PD patients | Up to 36 months
  The presence of genetic variations in the AQP4 gene, measured with single nucleotide polymorphisms will be correlated, in idiopathic and familial PD patients, with higher (worse) scores on the Hoehn & Yahr scales
Association between genetic variations in the AQP4 gene and worse cognitive symptoms in PD patients | Up to 36 months
  The presence of genetic variations in the AQP4 gene, measured with single nucleotide polymorphisms will be correlated, in idiopathic and familial PD patients, with lower (worse) scores on Montreal Cognitive Assessment (MoCA) scale
Association between genetic variations in the AQP4 gene and worse sleep symptoms in PD patients | Up to 36 months
  The presence of genetic variations in the AQP4 gene, measured with single nucleotide polymorphisms will be correlated, in idiopathic and familial PD patients, with worse sleep performances as assessed with sleep scales and Actigraph
Association between genetic variations in the AQP4 gene and worse non-motor symptoms in PD patients | Up to 36 months
  The presence of genetic variations in the AQP4 gene, measured with single nucleotide polymorphisms will be correlated, in idiopathic and familial PD patients, with higher (worse) scores on scales for non-motor symptoms.

SECONDARY OUTCOMES:
Association between genetic variations in the AQP4 gene and altered levels of glymphatic system markers in PD patients | Up to completion of study
  The presence of genetic variations in the AQP4 gene, measured with single nucleotide polymorphisms will be correlated, in idiopathic and familial PD patients, with increased levels of blood concentration of LRP-1, ABCB1 and AQP4
Association between genetic variations in the AQP4 gene and altered levels of astrocytic | Up to completion of study
  The presence of genetic variations in the AQP4 gene, measured with single nucleotide polymorphisms will be correlated, in idiopathic and familial PD patients, with increased levels of blood concentration of S100β
Association between genetic variations in the AQP4 gene and altered levels of protein aggregation markers in PD patients | Up to completion of study
  The presence of genetic variations in the AQP4 gene, measured with single nucleotide polymorphisms will be correlated, in idiopathic and familial PD patients, with increased levels of blood concentration of α-synuclein

CONTACTS AND LOCATIONS:
Overall Officials: Marios Politis, MD MSc PhD, Study Chair — University of Exeter
Locations (4):
- United Kingdom (4):
  - East Kent University Hospitals NHS Foundation Trust, Ashford
  - University of Exeter, Exeter
  - Prince Phillip Hospital, Llanelli
  - Lewisham and Greenwich NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers.